CLINICAL TRIAL: NCT00076427
Title: Evaluation of Clinical, Virologic and Immunologic Factors That Contribute to the Pathogenesis of Chronic Hepatitis C and Its Complications
Brief Title: Leukapheresis for Research on HCV-Coinfected Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040086; 04-I-0086
Record Dates: First submitted 2004-01-21; First posted 2004-01-22 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2015-06-09

CONDITIONS: Hepatitis C; HIV Infections
Keywords: Immunity; Liver; Apheresis; Cytokine; Virology; Hepatitis C; HCV; Hepatitis C co-infection
MeSH Terms: conditions — Hepatitis C; HIV Infections

SUMMARY:
This study will collect quantities of white blood cells from patients infected with the hepatitis C virus (HCV) for research on the interactions between HCV and the human immunodeficiency virus (HIV) in people infected with both of these agents. Several studies have shown that infection with HIV adversely affects liver disease due to HCV.

Patients 18 years of age and older who are infected with both HCV and HIV or with HCV alone may be eligible for this study. Candidates must not have liver failure and must not be undergoing treatment for HCV at the time of enrollment.

Participants will undergo leukapheresis to collect white blood cells. This procedure allows collection of larger numbers of cells than would be possible with simple blood drawing. For the procedure, blood is removed through a needle in the vein of one arm and spun in a machine that separates the blood into its components. The white cells are extracted and the rest of the blood is re-infused through the same needle or through a needle in the other arm. The procedure takes approximately 1-3 hours, depending on the amount of white cells being collected. A maximum of three leukapheresis procedures are done. If additional procedures are required, the patient will sign a new consent form. Procedures will be limited to no more than three times a year, or once every 4 months.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) and Hepatitis B (HBV) infection are known to cause morbidity and mortality especially among those who are coinfected with Human Immunodeficiency virus (HIV). HCV infected individuals who are also coinfected with HIV have more rapid progression of liver disease, abnormal diagnostic serologies, higher levels of HCV viremia, and markedly lower levels of therapeutic responses to the standard combination therapy with peginterferon and ribavirin.

The underlying immunopathogenesis of HCV and HBV infection, progression of liver disease, and interactions with HIV are not yet clearly understood. A clear understanding of the immune correlates of protection against HCV and HBV are important in development of a vaccine for HCV and novel immune-based therapeutics for the cure of HBV.

This study will recruit individuals who are coinfected with HIV and HCV and/or HBV as well as those who are monoinfected with HCV or HBV. The study will enroll 2 groups. Participants in the first group (hereafter referred to as Group 1) will consist of participants recruited for research and clinical related blood draws, leukapheresis, and liver biopsies for long term study participation. Participants in the second group (hereafter referred to as Group 2) will consist of participants with known or suspected HCV and/or HBV who need assistance with diagnosis or treatment.

Participants in Group 1 will be apheresed or undergo blood draw several times after enrollment and may be followed for up to 10 years. Participants in Group 2 will be evaluated for HBV and/or HCV infection or complications, or receive treatment. The expectation is that may be followed for one year.

Leukapheresis is used in Group 1 in order to obtain sufficient cells to pursue the following objectives: delineating B cell response to CD4+ T cell help, delineating CD8+ T factors associated with suppression of viral replication and normalization of immune function, characterizing natural killer function relative to HCV and/or HBV disease, and identifying biomarkers for progression of liver disease. The required number of mononuclear cells needed to perform these experiments can be easily and safely obtained using leukapheresis procedures in the Clinical Center Apheresis Unit. Participants who do not meet apheresis criteria may participate through routine blood draws to contribute to this research. All participants in Group 1 may also receive a liver biopsy at NIH (every 3 years for HIV/HCV coinfected and all HBV infected and every 5 years for HCV monoinfected subjects) to assess the progression of liver disease.

Treatment plans for Group 2 HBV and/or HCV will be in accordance with standard medical practice, and the number and length of additional visits and diagnostic evaluations will vary accordingly.

ELIGIBILITY:
* INCLUSION CRITERIA FOR BOTH GROUPS:
* Adult (18 years old or older)
* Either monoinfected with HCV or coinfected with HCV and HIV
* Willingness to give informed consent.
* Willing to undergo genetic testing
* Willing to have samples stored for future research.
* Must have a referring physician or clinic that will continue to provide medical care.

Note: An HCV/HIV coinfected individual is defined as any individual with all the following: 1) Positive ELISA and western blot test for HIV, and 2) Positive serology and/or positive HCV RNA test; An HCV monoinfected individual is defined as any individual with all of the following: 1) Positive serology and/or positive HCV RNA test, and 2) Negative ELISA test for HIV

INCLUSION CRITERIA FOR GROUP 1:

-Must be willing and able to make follow up visits for leukapheresis and blood draws at least once in the next 6 months

INCLUSION CRITERIA FOR GROUP 2:

-Must be referred by a physician for the purposes of confirming HCV diagnosis, complications from HCV, or standard HCV treatment management.

EXCLUSION CRITERIA FOR BOTH GROUPS

Have any other condition, which the investigator considers a contraindication to study participation.

EXCLUSION FOR GROUP 1:

* Evidence of liver failure on liver biopsy, abdominal ultrasound, or liver function blood tests
* Receiving HCV therapy at the time of enrollment
* Platelet count < 50,00 per mL
* Hematocrit < 28 percent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2004-01-14; Study Completion 2015-06-09

CONTACTS AND LOCATIONS:
Overall Officials: Colleen M Hadigan, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (4):
- United States (4):
  - Family and Medical Counseling Service, Washington D.C., District of Columbia
  - Unity Health Care/Walker Jones, Washington D.C., District of Columbia
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Gerlach JT, Diepolder HM, Jung MC, Gruener NH, Schraut WW, Zachoval R, Hoffmann R, Schirren CA, Santantonio T, Pape GR. Recurrence of hepatitis C virus after loss of virus-specific CD4(+) T-cell response in acute hepatitis C. Gastroenterology. 1999 Oct;117(4):933-41. doi: 10.1016/s0016-5085(99)70353-7. PMID 10500077
- [Background] Lechner F, Gruener NH, Urbani S, Uggeri J, Santantonio T, Kammer AR, Cerny A, Phillips R, Ferrari C, Pape GR, Klenerman P. CD8+ T lymphocyte responses are induced during acute hepatitis C virus infection but are not sustained. Eur J Immunol. 2000 Sep;30(9):2479-87. doi: 10.1002/1521-4141(200009)30:93.0.CO;2-B. PMID 11009080
- [Background] Thursz M, Yallop R, Goldin R, Trepo C, Thomas HC. Influence of MHC class II genotype on outcome of infection with hepatitis C virus. The HENCORE group. Hepatitis C European Network for Cooperative Research. Lancet. 1999 Dec 18-25;354(9196):2119-24. doi: 10.1016/s0140-6736(99)91443-5. PMID 10609818